CLINICAL TRIAL: NCT06501677
Title: Using Ecological Momentary Data to Inform a Web-intervention for Romantic Partners Concerned About Their Loved Ones Drinking
Brief Title: Using EMA Data to Inform a Web-intervention for Couples Concerned About Drinking
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Portland State University (Other)
Responsible Party: Principal Investigator, Karen Osilla, Principal Investigator, Stanford University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 71858
Record Dates: First submitted 2024-07-09; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Alcohol; Use, Problem
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Identify CP communication behaviors that elicit or inhibit DP drinking using EMA (No Intervention): Couples (N=50 dyads) with one CP and one DP will be recruited from social media. Both partners will independently complete baseline and follow-up surveys. Both the CP and DP will independently complete a 21-day EMA with three daily reports on their communication and DP's drinking (craving, motives, consumption, problems). We will identify specific CP communication behaviors as proximal and long-term predictors of the DP's drinking and non-drinking.
  Hyp1: CP punishing drinking (e.g., yelling) will relate to increases in DP drinking.
  Hyp2: CP rewarding drinking (e.g., bringing alcohol home) will relate to increases in DP drinking.
  Hyp3: CP rewarding sobriety (e.g., planning non-drinking activities) will relate to decreases in DP drinking.
- Develop and evaluate the feasibility and acceptability of a WBI providing personalized feedback (Experimental): We will use the Behavioral Intervention Technology Model framework to iteratively develop a four-session WBI that includes CRAFT principles and education about communication patterns learned in Aim 1. During the WBI, CPs will receive personalized feedback based on their baseline data on how their communication may influence their DP's drinking. We will evaluate the WBI's feasibility and acceptability with 15 CPs to iteratively improve the WBI.
  Interventions: Behavioral: WBI
- Perform a pilot randomized controlled trial (RCT) comparing WBI to psychoeducation control (Active Comparator): Outcomes include DP drinking (primary), CP well-being (e.g., depression, anxiety, social support), and relationship functioning (e.g., relationship distress). Although the WBI will target CPs, we will collect data from both partners (N=80 couples) at baseline and 1-month follow-up to evaluate effects.
  Hyp4: DP, CP, and relationship outcomes will show greater improvement in the WBI compared to control.
  Interventions: Behavioral: WBI

INTERVENTIONS:
Behavioral: WBI — The WBI will comprise of four sessions focusing on CRAFT principles including: (1) self-care, (2) positive communication including ways to increase responsiveness to the DP (PPR; i.e., actively listening, showing understanding, expressing interest in what their DP is thinking and feeling, and trying to see where the DPs is coming from), (3) understanding the DP's drinking reinforcers, and (4) supporting the DP if they want help and engaging in positive, healthy activities with the DP. ' partner.
  Each module will take ~20-30 minutes and each session will: (1) instill optimism in CPs, (2) be solution-focused, (3) emphasize that the CP is not responsible for the DP's behaviors, and (4) use a nonjudgmental, non-confrontational, empathetic style. The WBI intervention is focused on reduced drinking in the DP and improved CP wellness.
  Other Names: Partners Connect
  Arms: Develop and evaluate the feasibility and acceptability of a WBI providing personalized feedback; Perform a pilot randomized controlled trial (RCT) comparing WBI to psychoeducation control

SUMMARY:
Alcohol misuse is a prevalent and serious problem with significant harms to society, individuals, and their relationships. Romantic partners have a strong influence on their partner's behavior, uniquely positioning them as a motivator and supportive factor in changing their partner's alcohol use, but little evidence exists on the specific ways they can influence their partner. The impact this has on the quality of their relationship, communication, and overall well-being has yet to be explored. Thus, this study utilizes qualitative, quantitative, and ecological momentary assessment (EMA) data from both partners to develop a web-based intervention that applies communication-based personalized feedback to support the concerned partner (CP) in motivating their drinking partner (DP) to reduce drinking and other adverse relationship outcomes.

DETAILED DESCRIPTION:
Previous research by our team and others has shown that certain CP responses to their DP's drinking (e.g., using punishment such as expressing anger or sarcasm, or threatening to leave) lead to increased DP drinking and poorer relationship functioning. Effective CP communication may affect fluctuations in DP drinking, but its mechanism is poorly understood. Limitations of prior research include long intervals between data collection points and lack of real-time dyadic data.The proposed project will use EMA and dyadic data to identify specific CP behaviors that elicit and/or inhibit DP drinking which will directly inform a CP-focused intervention. CP-focused interventions, such as Community Reinforcement and Family Therapy (CRAFT), encourage CP positive communication and reinforcement as important tools in promoting the DP's treatment entry. The DPs of CPs receiving CRAFT are 2-3 times more likely to enter alcohol treatment compared with Al-Anon or Johnson interventions and CRAFT is also effective in improving CP mental health and relationship functioning. However, CRAFT is time- and resource-intensive (i.e., 12 in-person sessions), limiting access for CPs who lack time or are hesitant to seek help. The proposed study aims to adapt CRAFT as a new WBI developed for a community sample of CPs. In contrast to the goals of CRAFT that focus on DP treatment entry, our WBI goals focus on outcomes that may be more proximal to treatment initiation and more attainable with a WBI including improved DP drinking, CP mental health and relationship functioning. In doing so, we also target DPs with a continuum of drinking severity including those who may not need treatment. Using EMA findings that elucidate communication strategies that influence DP drinking, the WBI will include psychoeducation on interaction patterns commonly associated with DP drinking and personalized feedback based on CP baseline data to support changes in CP communication strategies. This research addresses an important problem of mitigating the adverse impact of alcohol misuse on individuals and their families. The expected outcome of this research is to leverage CP influence into an accessible, theoretically-informed intervention that will help CPs more effectively communicate with their DP for improvements to their DP's drinking behavior, their own well-being, and their relationship functioning.

ELIGIBILITY:
Concerned Partners:

Inclusion Criteria:

* be at least 18 years of age
* be in a romantic relationship
* live with their partner
* have a computer, tablet, or phone with internet access
* have no plans to separate from partner in next 60 days
* feel safe from partner violence

Exclusion Criteria:

* report 4/5+ on the AUDIT-C

Drinking Partners:

Inclusion Criteria:

* be at least 18 years of age
* report 4/5+ on the AUDIT-C
* have a computer, tablet, or phone with internet access
* feel safe from partner violence

Exclusion Criteria:

* in current treatment for alcohol
* concern about their CPs drinking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
DP Alcohol Use | Baseline, Daily (EMA), 1-month-follow-up
  The frequency of and amount of alcohol use, craving, and consequences experienced by the drinking partner
CP Well-Being | Baseline, 1-month-follow-up
  The severity of depression and anxiety symptoms, level of anger, and perceived social support in the concerned partner
CP-DP Relationship Quality | Baseline, Daily (EMA), 1-month-follow-up
  The degree of conflict and cohesion, style of communication, satisfaction, frequency of disagreement, and overall quality of the relationship

SECONDARY OUTCOMES:
CP Communication and Responsiveness about Drinking | Baseline, Daily (EMA), 1-month-follow-up
  The degree to which the concerned partner employs strategies to reduce the drinking partner's drinking and the level of enablement and responsiveness towards their drinking

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States